CLINICAL TRIAL: NCT06396884
Title: Continuous Non-Invasive Blood Pressure Monitoring Versus Intermittent During Spinal Anesthesia in Elderly Patients With Femoral Fracture: Observational Cohort Study
Brief Title: Hemodynamic Optimization During Spinal Anesthesia in the Elderly
Acronym: HORSE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5924
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-04

CONDITIONS: Non Invasive Hemodynamic Monitoring; Proximal Femur Fracture; Fluid Therapy
MeSH Terms: conditions — Proximal Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control Group: Elderly patients over 65 years of age who underwent surgery for femoral fracture under spinal anesthesia. These patients underwent oscillometric intermittent (5 mins) noninvasive blood pressure monitoring during the surgical procedure and received intraoperative hemodynamic management based on a liberal fluid therapy protocol.
  Interventions: Device: Oscillometric intermittent non-invasive blood pressure
- ClearSight Group: Elderly patients over 65 years of age who will undergo surgery for femoral fracture under spinal anesthesia. These patients will undergo continuous and non-invasive blood pressure monitoring using the ClearSight system, and fluid management according to a hemodynamic optimization protocol based on goal-directed fluid therapy
  Interventions: Device: ClearSight

INTERVENTIONS:
Device: Oscillometric intermittent non-invasive blood pressure — The hemodynamic management followed liberal fluid therapy, as determined by the attending anesthetist's discretion
  Groups: Control Group
Device: ClearSight — The hemodynamic management will be conducted in accordance to a goal-directed fluid therapy (GDFT) utilizing the Clearsight system monitoring.
  Groups: ClearSight Group

SUMMARY:
In elderly patients over 65 years of age, proximal femur fracture is the most common type of fracture, and surgical intervention is typically required for the majority of cases. Subarachnoid anesthesia is commonly used for this type of surgery. The objective of this study is to assess the efficacy of continuous non-invasive blood pressure and hemodynamic monitoring compared to traditional methods of blood pressure measurement in reducing the duration of hospitalization and the incidence of post-operative complications in elderly patients undergoing surgery for femur fracture under subarachnoid anesthesia.

DETAILED DESCRIPTION:
The proximal femoral fracture is the most frequent fracture in elderly patients over 65 years old, often affected by multiple comorbidities. It is one of the main causes of hospitalization in this population and is associated with high mortality rates.

Surgical treatment is indicated for the majority of fractures, and spinal anesthesia is the most commonly used technique for this type of surgery.

Hypotension is a very common side effect after spinal anesthesia, with a reported incidence of 16%-33%, attributable to a reduction in systemic vascular resistance, cardiac output, or both mechanisms. Several studies have demonstrated the association between intraoperative hypotension, usually defined as a mean arterial pressure <65 mmHg, myocardial and renal organ damage, and 30-day mortality.

In clinical practice oscillometric, non-invasive blood pressure measurement (NIBP) is the first choice of blood pressure monitoring in the majority of low and moderate risk surgeries. This monitoring system is a non-invasive cuff around the upper arm (NIBP-arm), which allows for non-invasive detection of blood pressure values, usually every 5 minutes.

New continuous noninvasive devices to acquire instantaneous arterial blood pressure (ClearSight™, Edwards) may be more sensitive to detect procedural hypotension. Additionally, this system provides advanced hemodynamic parameters not available with traditional oscillometric methods of blood pressure measurement, supporting the anesthesiologist in proactive hemodynamic management of the patient.

Several systematic reviews have demonstrated the effectiveness of hemodynamic optimization protocols in reducing postoperative complications. Orthopedic surgical procedures, along with abdominal and neurosurgical procedures, are among those that benefit most from the adoption of an advanced hemodynamic monitoring system associated with a Goal-Directed Therapy (GDT) protocol.

One hundred forty-six patients, aged ≥ 65 years, with an American Society of Anaesthesiologists' (ASA) score I-III, undergoing surgical intervention due to femoral fracture and spinal anaesthesia will be enrolled. Seventy-three patients from a prospectively enrolled cohort (ClearSight group) will be compared with seventy-three patients from a retrospective cohort (Control Group) who underwent the same type of surgery under spinal anesthesia between May 2023 and December 2023 and were included according to the same eligibility criteria.

In the retrospectively enrolled patient cohort (control group), an intermittent non-invasive blood pressure monitoring system was used, and intraoperative hemodynamic anesthetic management was not standardized but left to the discretion of the attending anesthesiologist, consistently with the protocols of the operating unit.

In the prospectively enrolled patient cohort (Clearsight group), continuous non-invasive monitoring of arterial pressure will be conducted using the ClearSight system, allowing clinicians to implement Goal-Directed Fluid Therapy.

The purpose of this study is to evaluate the effectiveness of continuous non-invasive blood pressure and hemodynamic monitoring compared to traditional methods of blood pressure detection in reducing length of hospital stay and the percentage of post-operative complications in elderly patients undergoing surgery for femoral fracture under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

Patients with American Society of Anesthesiologists (ASA) physical status I-III, candidate for surgical intervention for femoral fracture under spinal anesthesia.

Exclusion Criteria:

* Severe valvular heart disease
* Heart failure (New York Heart Association - NYHA class ≥ 3)
* Vascular system pathologies
* Allergy or hypersensitivity to local anesthetics
* Absolute contraindications to spinal anesthesia
* Patient refusal to participate to the study

Ages: 65 Years to 99 Years | Sex: All
Age Groups: Older Adult
Study Population: The study aims to enroll 146 patients aged over 65 years, with ASA (American Society of Anesthesiologists) scores I-III, undergoing surgery for femoral fracture under spinal anesthesia. After obtaining informed consent, 73 patients from a prospectively enrolled cohort (ClearSight group) will be compared with 73 patients from a retrospective cohort (Control Group) who underwent the same type of surgery under spinal anesthesia between May 2023 and December 2023 and were included based on the same eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of hospitalization | 10-15 days
  To compare the length of hospital stay among elderly patients undergoing surgery for femoral fractures under subarachnoid anesthesia, where continuous non-invasive blood pressure monitoring utilizing the ClearSight system is implemented along with a standardized protocol for hemodynamic optimization, with the duration of hospital stay observed in a retrospective cohort of patients undergoing similar surgery but with intermittent (every 5 minutes) non-invasive blood pressure monitoring not linked to a standardized protocol for hemodynamic optimization

SECONDARY OUTCOMES:
Incidence of at least one postoperative complication | 10-15 days
  To compare the incidence of at least one of the following postoperative complications: pneumonia, pulmonary edema, ARDS (acute respiratory distress syndrome), pulmonary embolism, deep vein thrombosis, myocardial infarction, arrythmias, AKI (acute kidney injury), surgical site infection, wound dehiscence, urinary tract infection, sepsis, paralytic ileus, diarrhea, acute cerebrovascular accidents, delirium

CONTACTS AND LOCATIONS:
Overall Officials: ROSSANO RF FESTA, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Rossano Festa, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jessen MK, Vallentin MF, Holmberg MJ, Bolther M, Hansen FB, Holst JM, Magnussen A, Hansen NS, Johannsen CM, Enevoldsen J, Jensen TH, Roessler LL, Lind PC, Klitholm MP, Eggertsen MA, Caap P, Boye C, Dabrowski KM, Vormfenne L, Hoybye M, Henriksen J, Karlsson CM, Balleby IR, Rasmussen MS, Paelestik K, Granfeldt A, Andersen LW. Goal-directed haemodynamic therapy during general anaesthesia for noncardiac surgery: a systematic review and meta-analysis. Br J Anaesth. 2022 Mar;128(3):416-433. doi: 10.1016/j.bja.2021.10.046. Epub 2021 Dec 13. PMID 34916049
- [Background] Moppett IK, Rowlands M, Mannings A, Moran CG, Wiles MD; NOTTS Investigators. LiDCO-based fluid management in patients undergoing hip fracture surgery under spinal anaesthesia: a randomized trial and systematic review. Br J Anaesth. 2015 Mar;114(3):444-59. doi: 10.1093/bja/aeu386. Epub 2014 Dec 11. PMID 25500940
- [Background] Lorente JV, Reguant F, Arnau A, Borderas M, Prieto JC, Torrallardona J, Carrasco L, Solano P, Perez I, Farre C, Jimenez I, Ripolles-Melchor J, Monge MI, Bosch J. Effect of goal-directed haemodynamic therapy guided by non-invasive monitoring on perioperative complications in elderly hip fracture patients within an enhanced recovery pathway. Perioper Med (Lond). 2022 Aug 10;11(1):46. doi: 10.1186/s13741-022-00277-w. PMID 35945605
- [Background] Brauer CA, Coca-Perraillon M, Cutler DM, Rosen AB. Incidence and mortality of hip fractures in the United States. JAMA. 2009 Oct 14;302(14):1573-9. doi: 10.1001/jama.2009.1462. PMID 19826027
- [Background] Kannegaard PN, van der Mark S, Eiken P, Abrahamsen B. Excess mortality in men compared with women following a hip fracture. National analysis of comedications, comorbidity and survival. Age Ageing. 2010 Mar;39(2):203-9. doi: 10.1093/ageing/afp221. Epub 2010 Jan 14. PMID 20075035
- [Background] Longo UG, Vigano M, de Girolamo L, Banfi G, Salvatore G, Denaro V. Epidemiology and Management of Proximal Femoral Fractures in Italy between 2001 and 2016 in Older Adults: Analysis of the National Discharge Registry. Int J Environ Res Public Health. 2022 Dec 17;19(24):16985. doi: 10.3390/ijerph192416985. PMID 36554865
- [Background] Carpenter RL, Caplan RA, Brown DL, Stephenson C, Wu R. Incidence and risk factors for side effects of spinal anesthesia. Anesthesiology. 1992 Jun;76(6):906-16. doi: 10.1097/00000542-199206000-00006. PMID 1599111
- [Background] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Background] Ahuja S, Mascha EJ, Yang D, Maheshwari K, Cohen B, Khanna AK, Ruetzler K, Turan A, Sessler DI. Associations of Intraoperative Radial Arterial Systolic, Diastolic, Mean, and Pulse Pressures with Myocardial and Acute Kidney Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2020 Feb;132(2):291-306. doi: 10.1097/ALN.0000000000003048. PMID 31939844
- [Background] Giglio M, Biancofiore G, Corriero A, Romagnoli S, Tritapepe L, Brienza N, Puntillo F. Perioperative goal-directed therapy and postoperative complications in different kind of surgical procedures: an updated meta-analysis. J Anesth Analg Crit Care. 2021 Dec 15;1(1):26. doi: 10.1186/s44158-021-00026-3. PMID 37386648